CLINICAL TRIAL: NCT06795724
Title: Effect of PENG Block on Inflammatory Parameters and Mortality in Geriatric Patients Undergoing Hip Fracture Surgery
Brief Title: Effect of Peng Block Application on Inflammation and Mortality in Hip Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Burak NALBANT, assistant professor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: E2-24-8891
Record Dates: First submitted 2025-01-16; First posted 2025-01-28 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Inflammatory Response; Anesthesia; Hip Fractures
Keywords: PENG block; inflammation; SIRI; Mortality; Hip fracture
MeSH Terms: conditions — Hip Fractures; Inflammation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG Block (Active Comparator): PENG block will be performed before the surgery. For PENG block, patients are in the supine position is deposited. The convex ultrasound probe is initially placed over the anterior superior iliac spine, then the probe moves medially until the femoral artery is visualized. In this view, iliopectineal eminence (IPE), iliopsoas muscle and tendon, femoral artery and iliac muscle are observed. Between the psoas tendon and the IPE 22 gauge 80 mm block needle is guided and 20cc local anesthetic used in % 0.25 bupivacaine is administered by intermittent aspiration.
  Interventions: Other: PENG block
- Control (Other): Standard analgesia method will be applied and analgesia will be provided with tramadol hydrochloride and paracetamol.
  Interventions: Other: Control

INTERVENTIONS:
Other: PENG block — For PENG block, patients are in the supine position is deposited. The convex ultrasound probe is initially placed over the anterior superior iliac spine, then the probe moves medially until the femoral artery is visualized. In this view, iliopectineal eminence (IPE), iliopsoas muscle and tendon, femoral artery and iliac muscle are observed. Between the psoas tendon and the IPE 22 gauge 80 mm block needle is guided and 20cc local anesthetic used in % 0.25 bupivacaine is administered by intermittent aspiration.
  Arms: PENG Block
Other: Control — Standard analgesia method will be applied and analgesia will be provided with tramadol hydrochloride and paracetamol.
  Arms: Control

SUMMARY:
In this study, the investigators the effect of PENG block on SIRI (systemic inflammation response index) and 30-day mortality in geriatric patients(over 65 years old) undergoing hip surgery, and the effect on the length of hospital stay.

DETAILED DESCRIPTION:
Patients over the age of 65 who were scheduled for surgery due to hip fracture were included in the study. According to the power analysis, it was estimated that at least 52 patients would be required for adequate statistical power. Initially, a total of 60 patients were assessed for eligibility and planned to be divided into two groups by randomization. Multimodal analgesia was applied to both groups.

The first group (Group P) received a preoperative Pericapsular Nerve Group (PENG) block, while the second group (Group C) did not receive an analgesic block and was given paracetamol and tramadol hydrochloride for analgesia. All patients received spinal anesthesia using 10 mg of hyperbaric bupivacaine.

Preoperatively, IL-6, CRP, and complete blood count (CBC) tests were performed on all patients, and these tests were repeated 4, 24, and 48 hours after the surgical stimulus. At the end of the operation, total blood loss, transfused blood products and their volumes, and operation time were recorded. Postoperatively, NRS pain scores, time to first analgesic requirement, length of hospital stay, and 30-day mortality were evaluated.

Post-Completion Study Flow

After completion of the study, a total of 60 patients were assessed for eligibility as planned. Of these, 2 patients declined to participate. The remaining 58 patients were randomized into two groups.

In Group P, one patient required conversion to general anesthesia during surgery. In Group C, two patients required intraoperative sedation, and one patient required conversion to general anesthesia. Therefore, four patients were excluded from the final analysis.

As a result, the analyses were conducted on 54 patients in total, with 28 patients in Group P and 26 patients in Group C.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2-3 score
* Hip Fracture Surgery

Exclusion Criteria:

* Refusal to participate in the study
* ASA score of 4 and above
* Obesity (BMI >40)
* Failure of spinal block
* Switching to general anesthesia
* Patients undergoing revision surgery
* Patients with multitrauma
* Patients with old fractures (>3 weeks)
* Patients receiving preoperative and intraoperative sedation
* Patients with active malignancy receiving RT, KT
* Patients with active infection, patients receiving antibiotic treatment
* Patients with contraindications for regional anesthesia techniques
* Patients receiving chronic treatment with steroids or immunosuppressants
* Patients using anti-inflammatory drugs

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2025-08-17 (Actual)

PRIMARY OUTCOMES:
SIRI-systemic inflammatory response index | Preoperative, Postsurgery 4. 24. 48.hour
  The systemic inflammatory response index (SIRI) is defined as "neutrophil count × monocytes/lymphocyte counts".
IL-6 | Preoperative, Postsurgery 4. 24. 48.hour
  Measurement of IL-6 level in blood

SECONDARY OUTCOMES:
CRP | Preoperative, Postsurgery 4. 24. 48.hour
  Measurement of CRP level in blood
SII | Preoperative, Postsurgery 4. 24. 48.hour
  systemic inflammation index (SII) is defined as "platelet count × neutrophil count/lymphocyte count"
NLR | Preoperative, Postsurgery 4. 24. 48.hour
  neutrophil-to-lymphocyte ratio
NRS score | Postoperative 0-2-8-16-24-36-48 hour
  The degree of pain will be measured with numerical rating scale (NRS). All patients' postoperative pain numerical rating scale (NRS-numeric rating scale; 0 = absence of pain, 10 = unbearable pain) will be recorded in both groups.
Additional analgesic requirement | Postoperative first 24 hour
  The time of first postoperative analgesic requirement will be noted.
length of hospital stay | 1 week
  total day of hospital stay will be noted
Mortality | Postoperative 30 day
  30-day mortality of patients will be followed.

CONTACTS AND LOCATIONS:
Overall Officials: burak nalbant, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fang Z, Gao B, Wang Z, Chen X, Liu M. Association of systemic inflammation response index with mortality risk in older patients with hip fracture: a 10-year retrospective cohort study. Front Med (Lausanne). 2024 May 22;11:1401443. doi: 10.3389/fmed.2024.1401443. eCollection 2024. PMID 38841577
- [Background] Gentili ME, Mazoit JX, Samii K K, Fletcher D. The effect of a sciatic nerve block on the development of inflammation in carrageenan injected rats. Anesth Analg. 1999 Oct;89(4):979-84. doi: 10.1097/00000539-199910000-00029. PMID 10512275